CLINICAL TRIAL: NCT06995508
Title: Managing Anorexia During Chemoradiation With Olanzapine (MACRO)
Brief Title: Olanzapine for Managing Anorexia in Head and Neck Cancer Patients Undergoing Chemoradiation, MACRO Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 3757323; NCI-2025-03335 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 3757323 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-05-12; First posted 2025-05-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cancer-Associated Anorexia; Head and Neck Squamous Cell Carcinoma; Neck Squamous Cell Carcinoma of Unknown Primary
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Practice Guidelines as Topic; Standard of Care; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (standard of care) (Active Comparator): Patients receive standard of care symptom management on study per the discretion of the treating institution.
  Interventions: Other: Best Practice; Other: Questionnaire Administration
- Arm II (olanzapine, standard of care) (Experimental): Starting day 1 of CRT, patients receive olanzapine PO QD for up to 10 weeks after completion of CRT in the absence of disease progression or unacceptable toxicity. Patients also receive standard of care symptom management on study per the discretion of the treating institution.
  Interventions: Other: Best Practice; Drug: Olanzapine; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Given standard of care symptom management
  Other Names: standard of care; standard therapy
Drug: Olanzapine — Given PO
  Other Names: LY 170053; Zyprexa; Zyprexa Zydis
  Arms: Arm II (olanzapine, standard of care)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial compares the effect of adding olanzapine to standard of care symptom management for nausea to standard of care alone in managing an abnormal loss of the appetite for food (anorexia) in patients treated with chemoradiation therapy (CRT) for head and neck cancer. Patients undergoing CRT may experience treatment-related side effects, including pain, nausea, and a discomfort in the ability to speak, swallow and eat. These side effects have been shown to increase weight loss, opiate use and hospitalization. Olanzapine is a drug used to treat certain mental disorders. It is also being studied in the treatment of nausea and vomiting caused by some cancer treatments. It is a type of anti-psychotic and a type of monoamine antagonist. Adding olanzapine to standard of care symptom management to limit nausea may be more effective than standard of care alone in managing anorexia in head and neck cancer patients during CRT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the effect of adding olanzapine to standard symptom management on preventing weight loss during chemoradiation.

SECONDARY OBJECTIVES:

I. To assess the effect of olanzapine on:

Ia. Preventing severe weight loss; Ib. The rate of toxicities possibly- or probably- related to the symptom management regimen;

Ic. Quality of Life (QOL) scores:

Ici. With particular attention to nausea, vomiting, appetite, loss, swallowing, pain; and Icii. Special attention to sleep; Id. Opiate use, hospitalization rate, feeding tube use, chemotherapy delays, and additional olanzapine prescriptions.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard of care symptom management on study per the discretion of the treating institution.

ARM II: Starting day 1 of CRT, patients receive olanzapine PO QD for up to 10 weeks after completion of CRT in the absence of disease progression or unacceptable toxicity. Patients also receive standard of care symptom management on study per the discretion of the treating institution.

After completion of study treatment, patients are followed up at 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Diagnosed with biopsy-proven, squamous cell carcinoma of the head and neck, including squamous cell carcinoma of the neck with unknown primary site
* Eligible for curative-intent chemoradiation therapy of the head and neck
* Patients must be eligible for concurrent systemic therapy (preferably platinum based) as determined by the treating medical oncologist to undergo platinum-based chemotherapy
* Ability to swallow and retain oral medication
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* While you are on study and taking olanzapine, you agree to avoid the following:

  * Taking the drug Symbyax (which already contains olanzapine)
  * Consuming alcohol
  * Operating hazardous machinery, including automobiles, until you are reasonably certain that the study drug therapy does not have any bad effects on your mental and physical health
* Participant must understand the investigational nature of this study and sign an institutional review board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Eligible for palliative-intent radiation therapy only
* Patients with a feeding tube
* Regular systemic steroid use
* Atypical antipsychotic use

  * Other dopamine receptor blockers routinely used as anti-emetics (eg. prochlorperazine/compazine and metoclopramide) are allowed to be prescribed as usual care on this study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, diabetes or psychiatric illness/social situations that would limit compliance with study requirements
* Known hypersensitivity to olanzapine
* Pregnant or nursing female participants
* Known history of seizures
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2030-11-15 (Estimated); Study Completion 2031-11-15 (Estimated)

PRIMARY OUTCOMES:
Average change in weight | From baseline to patient lowest weight during chemoradiation therapy (CRT) treatment, assessed up to 5 weeks after last dose of study treatment
  Will be summarized by study arm using the mean and standard deviation. A two-sample t-test will be used. All test assumptions will be verified graphically, and transformations or non-parametric approaches will be considered, as appropriate.

SECONDARY OUTCOMES:
Proportion of patients with severe weight loss | At baseline up to any time point during CRT treatment, assessed up to 5 weeks after last dose of study treatment
  Will be defined as >= 10% body weight loss. Will be summarized by study arm and compared by the Fisher exact test or chi-squared test as appropriate.
Incidence of adverse events | Up to 5 weeks after last dose of study treatment
  Will be assessed using the Cancer Therapy Evaluation Program National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Will be summarized by attribution and grade using frequencies and relative frequencies. Differences in CTCAE rates (grade 2 or higher) will be compared between groups using the Fisher exact Test or chi-Squared test as appropriate.
Change in quality of life (QOL) scores | Baseline up to 5 weeks after last dose of study treatment
  Will be assessed using the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) . The Oral Mucositis Weekly Questionnaire-Head and Neck Cancer will be used to describe the short-term effects of radiation on QOL during treatment. Scores will be assessed by comparing the within-patient change. The treatment effect will be estimated with a generalized linear mixed model, describing the continuous EORTC quality of life outcomes as a function of a random patient effect, and fixed effects for treatment assignment, time, the stratification factor, the treatment assignment and the treatment/time interaction. The magnitude, direction and 95% confidence interval for the adjusted interaction term estimate will be used to describe the effect of olanzapine in improving different QOL domains. An interaction p-value < 0.05 will be considered statistically significant.
Change in Quality of Life | Up to 5 weeks after last dose of study treatment
  Will be assessed using the EORTC QLQ-H&N43 module questionnaire. Mean change from
Changes in sleep | Baseline up to 5 weeks after last dose of study treatment
  Will be assessed using the Insomnia Severity Index (ISI) score and the ISI category. Differences between treatment arms for categorical or binary end points will be compared using the chi-square test or Fisher's exact test as appropriate. Differences between treatment arms for continuous variables will be compared using the Mann-Whitney U test. Differences between treatment arms for time-to-event end points will be compared using Kaplan-Meier estimates and the log-rank test.
Opiate use | Up to 5 weeks after last dose of study treatment
  Will be defined as proportion of patients requiring opiate prescription during CRT, time to first opiate in days, and total opiate use in morphine milligram equivalents. Differences between treatment arms for categorical or binary end points will be compared using the chi-square test or Fisher's exact test as appropriate. Differences between treatment arms for continuous variables will be compared using the Mann-Whitney U test. Differences between treatment arms for time-to-event end points will be compared using Kaplan-Meier estimates and the log-rank test.
Hospitalization rate | Up to 5 weeks after last dose of study treatment
  Will be defined as proportion of patients requiring inpatient hospital admission for any reason during CRT. Differences between treatment arms for categorical or binary end points will be compared using the chi-square test or Fisher's exact test as appropriate. Differences between treatment arms for continuous variables will be compared using the Mann-Whitney U test. Differences between treatment arms for time-to-event end points will be compared using Kaplan-Meier estimates and the log-rank test.
Feeding tube use | Up to 5 weeks after last dose of study treatment
  Will be defined as the proportion of patients requiring feeding tube insertion during CRT. Differences between treatment arms for categorical or binary end points will be compared using the chi-square test or Fisher's exact test as appropriate. Differences between treatment arms for continuous variables will be compared using the Mann-Whitney U test. Differences between treatment arms for time-to-event end points will be compared using Kaplan-Meier estimates and the log-rank test.
Chemotherapy delays | Up to 5 weeks after last dose of study treatment
  Will be defined as the proportion of patients requiring delays in chemotherapy during CRT. Differences between treatment arms for categorical or binary end points will be compared using the chi-square test or Fisher's exact test as appropriate. Differences between treatment arms for continuous variables will be compared using the Mann-Whitney U test. Differences between treatment arms for time-to-event end points will be compared using Kaplan-Meier estimates and the log-rank test.
Additional olanzapine prescriptions | Up to 5 weeks after last dose of study treatment
  Will be defined as the proportion of patients prescribed olanzapine for intractable nausea during CRT.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag K Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States